CLINICAL TRIAL: NCT01842451
Title: A Phase 2, Multicenter, Randomized, Partially-Blind, Dose-Ranging Study to Evaluate the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of VX-135 and Daclatasvir in Treatment-Naïve Adult Subjects With Genotype 1 Chronic Hepatitis C
Brief Title: A Phase 2 Study to Evaluate the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of VX-135 and Daclatasvir in Subjects With Genotype 1 Chronic Hepatitis C Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VX13-135-105
Record Dates: First submitted 2013-04-24; First posted 2013-04-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Hepatitis C; CHC; HCV; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — daclatasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VX-135 High Dose with Daclatasvir (Experimental): 12 weeks of a high dose of VX-135 in combination with Daclatasvir
  Interventions: Drug: VX-135; Drug: Daclatasvir
- VX-135 Low Dose with Daclatasvir (Experimental): 12 weeks of a low dose of VX-135 in combination with Daclatasvir
  Interventions: Drug: VX-135; Drug: Daclatasvir

INTERVENTIONS:
Drug: VX-135
Drug: Daclatasvir

SUMMARY:
A Phase 2 Study to Evaluate the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of VX-135 and Daclatasvir in Treatment-Naïve Adult Subjects With Genotype 1 Chronic Hepatitis C

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have genotype 1 CHC and evidence of HCV infection at least 6 months before screening
* Subjects must be treatment-naïve and have not received prior treatment with any interferon, immunomodulatory agent, or DAA for HCV

Exclusion Criteria:

* Evidence of cirrhosis
* History or other clinical evidence of significant or unstable cardiac disease
* Any other cause of significant liver disease in addition to hepatitis C
* Creatinine clearance ≤50 mL/min using the Cockcroft-Gault equation at screening
* Female subjects who are pregnant or nursing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability as assessed by adverse events (AEs), vital signs, 12-lead electrocardiograms (ECGs), echocardiograms, and laboratory assessments | Up to 64 weeks

SECONDARY OUTCOMES:
The proportion of subjects who have a sustained virologic response (SVR; i.e., HCV RNA concentration below the lower limit of quantitation [<LLOQ; <25 IU/mL]) at 4 weeks after the last planned dose of treatment (SVR4) | Up to 20 Weeks
The proportion of subjects who have an SVR at 12 weeks after the last planned dose of treatment (SVR12) | Up to 28 weeks
The proportion of subjects who have an SVR at 44 weeks after the last planned dose of treatment (SVR24) | Up to 40 weeks
The proportion of subjects who have virologic relapse | Up to 64 weeks
The proportion of subjects who have virologic breakthrough | Up to 16 weeks
The amino acid sequence of the nonstructural NS5A and NS5B proteins in subjects who have treatment failure | Up to 64 weeks
The proportion of subjects who achieve SVR12 by HCV genotype 1 subtype (1a versus non-1a) | Up to 28 weeks
The proportion of subjects who achieve SVR12 by IL-28B genotype (CC versus non-CC) | Up to 28 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - New Zealand, Auckland
  - New Zealand, Christchurch